CLINICAL TRIAL: NCT03672916
Title: Allofit® IT Ceramic Bearing System in Total Hip Arthroplasty: A Multi-center, Prospective, Non-controlled Post Market Surveillance Study
Brief Title: Allofit® IT Ceramic Bearing System in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2010-24H
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Avascular Necrosis of Hip; Osteoarthritis, Hip; Inflammatory Arthritis; Post-Traumatic Osteoarthritis of Hip
Keywords: Total hip arthroplasty; Medical Device; Safety; Hip prosthesis
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients who received the Allofit IT with BIOLOX delta: Subjects in need of a primary total hip arthroplasty, who met the inclusion/exclusion criteria and who received the Allofit IT Shell in combination with the BIOLOX delta Taper Liners

SUMMARY:
This is a multi-center, prospective, non-controlled post market surveillance study. The objectives of this study are to obtain survival and outcome data on the Allofit IT Shell in combination with the BIOLOX® delta Taper Liner when used in primary total hip arthroplasty.

DETAILED DESCRIPTION:
The objectives of this study are to obtain survival and outcome data on the Allofit IT Shell in combination with the BIOLOX® delta Taper Liner when used in primary total hip arthroplasty.

This will be done by analysis of standard scoring systems, radiographs and adverse event records. Data will be used to monitor pain, mobility and survivorship, and to confirm the safety and performance of the Allofit IT Ceramic Bearing System.

A total of 200 patients are planned to be enrolled in this study which will last 12 years (2 year enrollment plus 10 years follow-up) with the follow-up visits at 6 months, 1, 2, 3, 5, 7, and 10 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 75 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN)
  * Osteoarthritis (OA)
  * Inflammatory arthritis (i.e. Rheumatoid arthritis)
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) of the affected hip joint(s).
* Patient has a Harris Hip Score <70 in the affected hip
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant.
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has a vascular (large and small vessel disease) insufficiency.
* The patient has a neurologic condition in the ipsalateral or contralateral limb which affects lower limb function.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give informed consent, or to comply with the follow-up program.
* The patient has received an investigational drug or device within the previous 6 months.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has osteoradionecrosis in the operative hip joint
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.
* The patient has known local bone tumors in the operative hip.
* The patient is Grade III obese with a Body Mass Index (BMI) > 40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of a maximum of 200 males and females who require primary total hip arthroplasty. Subjects will be enrolled at 4 investigative centers. Subjects must be geographically accessible throughout the study and be willing and able to attend required follow-up appointments. Candidates who express interest in study participation will be offered informed consent, and eligibility will be determined based upon the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (4):
- Germany (3):
  - Sana Kliniken Sommerfeld, Kremmen
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - LVR-Klinik für Orthopädie, Viersen
- Skåne University Hospital, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Started | 185
Completed | 133
Not Completed | 52
Not completed — Death | 6
Not completed — Lost to Follow-up | 29
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: Age (years) at date of surgery] | 56.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 48
  Germany | 136

OUTCOME MEASURES:

1. Primary Outcome: Survivorship
Description: The objective of this study is implant survival at 10 years which is assessed by revision of the the study device calculated using the Kaplan-Meier Survival Estimation. The survivorship with Kaplan-Meier (K-M) was calculated at 10 year for endpoint revision of any component.
Time Frame: 10 years post-surgery
Population: All study patients
Measure: Number; unit: Implants
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
Implants | 179

2. Primary Outcome: Safety of the Implant
Description: Will be evaluated by monitoring the frequency and incidence of adverse events (AE), serious adverse events (SAE), adverse device effects (ADE) and serious adverse device effects (SADE) b) Efficacy:
Time Frame: Up to 10 years postoperative
Population: The count of all participants with adverse events is summarized. Details are available in the Adverse Event overview of the results section
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
Participants
  Hip Related complications (AE and SAE) | 9
  Revisions | 6
  SAE's not related to study hip | 38

3. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). To obtain a final score, the points are summed. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
score on a scale
  Pre-op | 48.8 (11.5)
  6 months: number analyzed (Participants) | 148
  6 months | 93.2 (11.3)
  1 Year: number analyzed (Participants) | 165
  1 Year | 96.1 (7.9)
  2 Year: number analyzed (Participants) | 149
  2 Year | 96.9 (6.9)
  3 Year: number analyzed (Participants) | 136
  3 Year | 96.1 (9)
  5 Year: number analyzed (Participants) | 138
  5 Year | 95.2 (9.5)
  7 Year: number analyzed (Participants) | 129
  7 Year | 96.0 (8.3)
  10 Year: number analyzed (Participants) | 127
  10 Year | 93.9 (11.3)

4. Secondary Outcome: EQ-5D
Description: The EQ-5D-3L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life. The questionnaire includes five dimensions referring to mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in three ways/levels indicating no problems, some problems, and extreme problems. In the derived EQ-5D-3L score, the highest score is 1 and the lowest score is -0.594; negative numbers correspond to a self-assessed health state worse than being dead.
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: The number of participants decreased over time, reasons are: questionnaire not completed in full (score calculation not possible), missed visits, lost to follow-up or withdrawn from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 184
score on a scale
  pre-op | 0.4 (0.3)
  6 months: number analyzed (Participants) | 148
  6 months | 0.9 (0.2)
  1 Year: number analyzed (Participants) | 160
  1 Year | 0.9 (0.2)
  2 Year: number analyzed (Participants) | 154
  2 Year | 0.9 (0.2)
  3 Year: number analyzed (Participants) | 139
  3 Year | 0.9 (0.2)
  5 Year: number analyzed (Participants) | 141
  5 Year | 0.8 (0.2)
  7 Year: number analyzed (Participants) | 129
  7 Year | 0.8 (0.2)
  10 Year: number analyzed (Participants) | 130
  10 Year | 0.8 (0.2)

5. Secondary Outcome: SF-12 Physical and Mental Functional Scores
Description: The SF-12 is a multipurpose short-form (SF) generic measure of health status. It consists of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Scores ranges from 0 to 100, with higher scores indicating better physical and mental health functioning and lower scores indicating worse physical and mental health functioning.
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
score on a scale
  Pre-op, SF12 Physical: number analyzed (Participants) | 172
  Pre-op, SF12 Physical | 28.8 (7.1)
  6 months, SF12 Physical: number analyzed (Participants) | 142
  6 months, SF12 Physical | 46.5 (9.9)
  1 Year, SF12 Physical: number analyzed (Participants) | 158
  1 Year, SF12 Physical | 48.5 (8.9)
  2 Year, SF12 Physical: number analyzed (Participants) | 143
  2 Year, SF12 Physical | 49.5 (9.3)
  3 Year, SF12 Physical: number analyzed (Participants) | 135
  3 Year, SF12 Physical | 47.0 (10.6)
  5 Year, SF12 Physical: number analyzed (Participants) | 140
  5 Year, SF12 Physical | 46.9 (9.8)
  7 Year, SF12 Physical: number analyzed (Participants) | 130
  7 Year, SF12 Physical | 47.2 (10.8)
  10 Year, SF12 Physical: number analyzed (Participants) | 130
  10 Year, SF12 Physical | 47.3 (9.9)
  Pre-op, SF12 Mental | 44.9 (11.8)
  6 months, SF12 Mental: number analyzed (Participants) | 149
  6 months, SF12 Mental | 55.7 (7.9)
  1 Year, SF12 Mental: number analyzed (Participants) | 162
  1 Year, SF12 Mental | 55.0 (7.8)
  2 Year, SF12 Mental: number analyzed (Participants) | 148
  2 Year, SF12 Mental | 55.6 (7.2)
  3 Year, SF12 Mental: number analyzed (Participants) | 137
  3 Year, SF12 Mental | 54.6 (8.4)
  5 Year, SF12 Mental: number analyzed (Participants) | 139
  5 Year, SF12 Mental | 54.1 (9.1)
  7 Year, SF12 Mental: number analyzed (Participants) | 130
  7 Year, SF12 Mental | 52.5 (10.4)
  10 Year, SF12 Mental: number analyzed (Participants) | 130
  10 Year, SF12 Mental | 54.2 (8.1)

6. Secondary Outcome: UCLA Activity Score
Description: The case administered University of California at Los Angeles (UCLA) score allows assessment of the case's activity level at each time point with scores from 1 (Wholly inactive: dependent on others; cannot leave residence) to 10 (Regularly participates in impact sports)
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: The number of participants decreased over time, reasons are: questionnaire not completed, missed visits, lost to follow-up or withdrawn from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
score on a scale
  Pre-op | 4.3 (1.6)
  6 months: number analyzed (Participants) | 152
  6 months | 6.1 (1.7)
  1 Year: number analyzed (Participants) | 165
  1 Year | 6.4 (1.5)
  2 Year: number analyzed (Participants) | 154
  2 Year | 6.6 (1.6)
  3 Year: number analyzed (Participants) | 139
  3 Year | 6.2 (1.7)
  5 Year: number analyzed (Participants) | 141
  5 Year | 6.4 (1.7)
  7 Year: number analyzed (Participants) | 130
  7 Year | 6.0 (1.9)
  10 Year: number analyzed (Participants) | 130
  10 Year | 6.4 (1.7)

7. Secondary Outcome: Radiographic Evaluations
Description: Radiographic evaluation was done to assess (radiolucency, osteolysis, subsidence, cup migration, change in cup angle and change in femoral shaft angle) of study subjects who received the Allofit IT Acetabular System
Time Frame: 10 Years post-surgery
Population: All study patients
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
Number analyzed (Participants) | 185
Participants
  Stem Subsidence (0.2mm - 6mm) | 11
  Radiolucency (>2mm) | 4
  Cup Migration (0.3mm - 0.9mm) | 6
  Osteolysis | 1
  Heterotopic Ossification (Class III and class IV) | 3
  Calcar Resorption (0.3mm - 5mm) | 9

ADVERSE EVENTS:
Time Frame: From surgery until the last study visit at 10 years post-op.
Description: ISO definitions are applicable
Arm/Group | Patients Who Received the Allofit IT With BIOLOX Delta
All-Cause Mortality (participants affected / at risk) | 6/185
Serious Adverse Events (participants affected / at risk) | 45/185
Other Adverse Events (participants affected / at risk) | 52/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Allofit IT With BIOLOX Delta (N=185)
Study-hip affected: Revisions of implant system (Surgical and medical procedures) | 6 (6) — One or more components revised. Reasons for revision: dislocation (N=4), femur fracture (N=1), deep infection (N=1)
Study-hip affected: Luxation/Dislocation (Surgical and medical procedures) | 2 (3)
Study-hip affected: Periprosthetic femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (non-study hip) (Musculoskeletal and connective tissue disorders) | 22 (26) — Includes contralateral THA, TKAs, etc
Cardiovascular (Cardiac disorders) | 10 (10)
Oncological (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Infection (non-study hip) (Infections and infestations) | 2 (2)
Neurological (Nervous system disorders) | 2 (2)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Reported deaths with unknown causes (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Allofit IT With BIOLOX Delta (N=185)
Study-hip affected adverse events (Musculoskeletal and connective tissue disorders) | 6 (6) — Squeaking hip (N=4), pain due to a fall (N=1), periprosthetic femur fracture (N=1)
Musculoskeletal (non-study hip) (Musculoskeletal and connective tissue disorders) | 28 (36) — Includes osteoarthritis other joints, fractures, pain, etc
Cardiovascular (Cardiac disorders) | 11 (11)
Oncological (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Infection (Infections and infestations) | 3 (3)
Endocrine (Endocrine disorders) | 3 (3)
Neurological (Nervous system disorders) | 2 (2)
Others (General disorders) | 5 (5) — Psychiatric disorder (N=2), Respiratory (N=1), Gastrointestinal (N=1), Dermatological (N=1),

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03672916/Prot_SAP_000.pdf